CLINICAL TRIAL: NCT07252206
Title: Culturally-adapted Cognitive-behavioural Therapy for Black Sub-Saharan African and Caribbean People Experiencing Psychosis: A Case Series
Brief Title: A Case Series of Culturally-adapted CBTp for Black People in the UK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Peter Panayi, Principal Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS002287
Record Dates: First submitted 2025-09-30; First posted 2025-11-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Psychosis; Schizophrenia Spectrum Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy (Experimental)
  Interventions: Behavioral: Culturally-adapted cognitive-behavioural therapy

INTERVENTIONS:
Behavioral: Culturally-adapted cognitive-behavioural therapy — Cognitive-behavioural therapy for psychosis culturally-adapted for Black Sub-Saharan African and Caribbean people using a dedicated, integrated treatment manual

SUMMARY:
The goal of this case series study is to learn if culturally-adapted cognitive-behavioural therapy is practical, acceptable and safe among Black Sub-Saharan African and Caribbean people experiencing psychosis. The main question it aims to answer is:

Is culturally-adapted CBT for psychosis feasible, acceptable to and safe for Black Sub-Saharan African and Caribbean people experiencing psychosis?

Participants will be asked to:

* Answer some questionnaires about how things are at the moment
* Attend up to 16 sessions of therapy
* Answer the same questionnaires to see what has changed, if anything
* Complete a semi-structured interview about their expectations and experience of therapy

ELIGIBILITY:
Inclusion Criteria:

* Service users who identify as Black British, Black Caribbean, Black African, African-Caribbean or Mixed African/Caribbean with at least one parent and/or grandparent born in a Sub-Saharan African or Caribbean country
* People with a current ICD-10 schizophrenia spectrum disorder diagnosis, or who are currently receiving or have received support from an Early Intervention in Psychosis team
* 16 years or older
* Sufficient understanding of English to complete study measures and engage with CBTp

Exclusion Criteria:

* Current, primary diagnosis of substance use disorder
* Organic aetiology of psychosis
* Lacking capacity to provide full informed consent
* Currently experiencing a mental health crisis (i.e., are open to a home-based treatment team; are currently under Section of the Mental Health Act or have been under Section in the past 3 months) or immediate high risk to self or others (i.e., current suicidal intent or plans; unmanaged and intense non-suicidal self-injury)
* Currently receiving CBTp or received CBTp within the preceding 3 months
* Unwilling to participate in culturally-adapted CBTp

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Semi-structured qualitative interview: Service user acceptability | End of therapy (16 weeks)
  Service user satisfaction as assessed by qualitative interview.

SECONDARY OUTCOMES:
Working Alliance Inventory-Short Form Revised | End of therapy (16 weeks)
  Acceptability measured sessionally using the Working Alliance Inventory-Short Form Revised (Hatcher & Gillaspy, 2006)
Adverse Events Checklist | Each therapy session (16 weeks)
  Safety monitored sessionally using an Adverse Events Checklist developed for this study
Subjective Experience of Psychosis Scale | End of therapy (16 weeks)
  Subjective distress measured by the Subjective Experience of Psychosis Scale (Haddock et al., 2011)
Questionnaire about the Process of Recovery | End of therapy (16 weeks)
  Perceived recovery measured by the Questionnaire about the Process of Recovery (Law et al., 2014)
Depression, Anxiety and Stress Scales | End of therapy (16 weeks)
  Emotional wellbeing measured by the Depression, Anxiety and Stress Scales (Lovibond & Lovibond, 1995)

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Manchester Mental Health NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No